CLINICAL TRIAL: NCT03064100
Title: Pilot Evaluation of the FilmArray® Childhood Systemic Infection (CSI) Panel
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: BioFire Diagnostics, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: BFDxCSIPilot
Record Dates: First submitted 2017-02-14; First posted 2017-02-24 (Actual); Last update posted 2017-07-21 (Actual); Status verified 2017-02

CONDITIONS: Systemic Infection
MeSH Terms: conditions — Toxemia | interventions — Observation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma and Whole Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Specimens that meet inclusion criteria
  Interventions: Other: Observational Study

INTERVENTIONS:
Other: Observational Study — Exclusion from the study

SUMMARY:
The purpose of this study is to collect data to support decisions made by BioFire regarding assay development, panel composition, and intended use for the final FilmArray CSI reagent pouch. The study will utilize whole blood and/or plasma obtained from pediatric patients under 18 years of age that present with acute fever.

ELIGIBILITY:
Inclusion Criteria:

* Subject has presented to the ED and is suspected of a systemic infection as indicated by a clinician order for blood culture
* Parent/guardian gives written permission (and assent is obtained from children of sufficient maturity)
* Blood specimen can be collected at the same time as the blood culture during the ED visit (or within 12 hours of being admitted from the ED)
* Specimen is at least 500 µL (1.5 mL collection desired)

Exclusion Criteria:

* Parent/guardian is unavailable or unable to give permission, or assent is not obtained (from children of sufficient maturity)
* Physician determines that participation in the study is an unacceptable health risk
* Minimum volume requirement is not met

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatric patients under the age of 18 suspected of systemic infection
Sampling Method: Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2017-03-21 (Actual); Primary Completion 2018-02 (Estimated); Study Completion 2018-02 (Estimated)

PRIMARY OUTCOMES:
Sensitivity (or positive percent agreement) and specificity (or negative percent agreement) of the assays comprising FilmArray CSI Panel with respect to reference methods (bacterial culture and independent molecular assays) | 12 months

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Children's Hospital of Los Angeles, Los Angeles, California
  - Emory University, Atlanta, Georgia
  - Children's Mercy Hospital, Kansas City, Missouri

IPD SHARING:
Plan to Share IPD: No